CLINICAL TRIAL: NCT02723006
Title: An Open-Label, Phase 1b, Multi-Arm Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of Investigational Treatments in Combination With Standard of Care Immune Checkpoint Inhibitors in Patients With Advanced Melanoma
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of Investigational Treatments in Combination With Standard of Care Immune Checkpoint Inhibitors in Participants With Advanced Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision: Protocol efficacy futility met
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C28003; U1111-1177-4142 (Other: WHO); 2015-005554-35 (EudraCT Number)
Record Dates: First submitted 2016-03-25; First posted 2016-03-30 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Melanoma
Keywords: Drug Therapy
MeSH Terms: conditions — Melanoma | interventions — tovorafenib; plozalizumab; vedolizumab; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TAK-580 + nivolumab (Experimental): TAK-580 orally, once weekly along with nivolumab, intravenous, every 2 weeks.
  Interventions: Drug: TAK-580; Drug: nivolumab
- TAK-202 (plozalizumab) + nivolumab (Experimental): TAK-202 (plozalizumab) 2 milligram (mg), intravenous, once in Week 1, 3, 5, 9, and every 4 weeks thereafter with nivolumab infusion, intravenous, every 2 weeks.
  Interventions: Drug: TAK-202; Drug: nivolumab
- vedolizumab + nivolumab + ipilimumab (Experimental): Vedolizumab intravenous, once in Week 1, 3, 5, and 13 along with nivolumab infusion, intravenous, once in Week 1, 4, 7, 10, and 13 and every 2 weeks thereafter, along with ipilimumab intravenous, once in Week 1, 4, 7, and 10.
  Interventions: Drug: vedolizumab; Drug: nivolumab; Drug: ipilimumab

INTERVENTIONS:
Drug: TAK-580 — TAK-580 tablets
  Other Names: MLN2480
  Arms: TAK-580 + nivolumab
Drug: TAK-202 — TAK-202 infusion
  Other Names: MLN1202; plozalizumab
  Arms: TAK-202 (plozalizumab) + nivolumab
Drug: vedolizumab — vedolizumab infusion
  Other Names: Entyvio
  Arms: vedolizumab + nivolumab + ipilimumab
Drug: nivolumab — nivolumab infusion
  Other Names: Opdivo
Drug: ipilimumab — ipilimumab infusion
  Other Names: Yervoy
  Arms: vedolizumab + nivolumab + ipilimumab

SUMMARY:
The purpose of this study is to determine the initial safety profile and initial antitumor activity of the combination treatments (immune checkpoint inhibitors [nivolumab, ipilimumab] with investigational drugs [TAK-580, TAK-202 (plozalizumab), vedolizumab]) in the 3 arms when administered to participants with advanced melanoma.

DETAILED DESCRIPTION:
The drugs being tested in this study are called TAK-580, TAK-202 (plozalizumab), and vedolizumab. These investigational drugs were given along with standard of care checkpoint inhibitors ([nivolumab in Arms 1 and 2] or nivolumab + ipilimumab in Arm 3). This study looked at the safety profile of the combination treatments in each arm when administered to participants with metastatic melanoma.

The study planned to enroll approximately 156 participants. Participants were assigned to one of the 3 treatment groups:

* TAK-580 + nivolumab
* TAK-202 (plozalizumab) + nivolumab
* vedolizumab + nivolumab + ipilimumab

This study consists of 3 parts. A dose-escalation safety lead-in phase, confirmatory safety phase and a cohort expansion phase. This multi-center trial will be conducted in the United States. The overall time to participate in this study is 50 weeks. Participants may make multiple visits to the clinic and 30, 60, and 90 days after last dose of study drug for follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or female participant of 18 years or older.
2. Has histologically confirmed, unresectable Stage III or Stage IV melanoma per the American Joint Committee on Cancer (AJCC) staging system.
3. Has an eastern cooperative oncology group (ECOG) performance status of 0-1.
4. Adequate bone marrow reserve and renal and hepatic function within 28 days before the first dose of study drug on the basis of the defined laboratory parameters.
5. For TAK-580 + nivolumab and TAK-202 (plozalizumab) + nivolumab only: Had disease accessible for repeat nonsignificant risk biopsy (those occurring outside the brain, lung/mediastinum, and pancreas, or obtained with endoscopic procedures extending beyond the esophagus, stomach, or bowel) and willingness to undergo serial tumor biopsies.
6. Additional Inclusion Requirements for TAK-580 + nivolumab

   a) BRAF V600 mutation-positive or NRAS mutation-positive disease previously untreated with RAF, MEK, or other inhibitors of the mitogen-activated protein kinase (MAPK) pathway. Participants who have progressed on these agents can still be enrolled in TAK-202 (plozalizumab) + nivolumab or vedolizumab + nivolumab + ipilimumab.
7. Additional Inclusion Requirements for expansion cohorts only a) Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (Version 1.1) and at least 1 nonsignificant risk, non-target lesion accessible for biopsy per the guidelines above (for TAK-580 + nivolumab and TAK-202 (plozalizumab) + nivolumab only).

Exclusion Criteria:

1. Has active brain metastases or leptomeningeal metastases. Participants with brain metastases are eligible if these have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for at least 4 weeks after treatment is complete and within 28 days prior to first dose of study drug administration. There must also be no requirement for high doses of systemic corticosteroids that could result in immunosuppression (greater than [>] 10 milligram per day [mg/day] prednisone equivalents) for at least 2 weeks prior to study drug administration.
2. Completed a prior therapy less than (<) 2 weeks prior to first dose and for whom adverse events (AEs) related to prior therapy had not returned to baseline or improved to Grade 1.
3. Has active, known or suspected autoimmune disease.
4. Has a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of study drug administration.
5. Has a history of pneumonitis requiring treatment with steroids; history of idiopathic pulmonary fibrosis (including pneumonitis), interstitial lung disease, drug-induced pneumonitis, organizing pneumonia, or evidence of active pneumonitis on screening chest computed tomography (CT) scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted.
6. Is previously diagnosed human immunodeficiency virus (HIV) infection or active hepatitis B or C.
7. Additional Exclusion Requirements for arm 1 only (nivolumab Plus TAK-580)

   1. Concomitant use or administration of clinically significant enzyme inducers less than or equal to (<=) 14 days before the first dose of TAK-580.
   2. Treatment with gemfibrozil (or other strong CYP2C8 inhibitor) within 14 days before the first dose of TAK-580.
   3. Left ventricular ejection fraction (LVEF) <50 percent (%) as measured by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA) within 4 weeks before receiving the first dose of study drug.
   4. Known gastrointestinal (GI) disease or prior GI procedure that could interfere with the oral absorption or tolerance of the TAK-580.
8. Additional Exclusion Requirements for arm 3 only (vedolizumab Plus nivolumab Plus ipilimumab)

   1. Had prior exposure to rituximab, natalizumab, vedolizumab, or alemtuzumab.
   2. Has a history of any major neurological disorders, including stroke, multiple sclerosis, or neurodegenerative disease.
   3. Has taken any live vaccinations within 30 days before study drug administration except for the influenza vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (14):
- United States (14):
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of California San Francisco Medical Center, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Emory University Hospital, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - New York University Langone Medical Center, New York, New York
  - Saint Luke's Cancer Center - Bethlehem, Easton, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Inova Fairfax Hospital, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: http://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 10 investigative sites in the United States from 22 June 2016 to 11 May 2018.
Pre-assignment Details: Participants with advanced/metastatic melanoma were enrolled to receive:TAK-580+nivolumab,TAK-202+nivolumab,or vedolizumab+nivolumab+ipilumab. Study was terminated early after the dose escalation safety-lead in phase due to lack of enrollment(Arm 1), lack of clinical benefit(Arm 2), and after pre-specified stopping rule for diarrhea was met(Arm 3).
Groups:
- Arm 1: TAK-580 + Nivolumab: Participants in this group received TAK-580 400 milligram (mg), tablets, orally, once weekly along with nivolumab 3 milligram per kilogram (mg/kg), infusion, intravenous, once every 2 weeks (up to Week 48).
- Arm 2: TAK-202 + Nivolumab: Participants in this group received TAK-202 (plozalizumab) 4 mg/kg titrated up to 8 mg/kg (stable dose), infusion, intravenous, once in Weeks 1, 3, 5, and every 4 weeks thereafter along with nivolumab 3 mg/kg, infusion, intravenously, once every 2 weeks (up to Week 50).
- Arm 3: Vedolizumab + Ipilimumab + Nivolumab: Participants in this group received vedolizumab 200 mg titrated up to 450 mg (stable dose), infusion, intravenously, once in Weeks 1, 3, 5, and 13 along with ipilimumab 3 mg/kg, infusion, intravenously, once every 3 weeks for 4 doses and nivolumab 1 mg/kg, infusion, intravenously, once every 3 weeks for 4 doses, followed by nivolumab 3 mg/kg, infusion, intravenously, once every 2 weeks until disease progression or unacceptable toxicity (up to Week 48).
Period: Overall Study
Arm/Group | Arm 1: TAK-580 + Nivolumab | Arm 2: TAK-202 + Nivolumab | Arm 3: Vedolizumab + Ipilimumab + Nivolumab
Started | 1 | 9 | 12
Completed | 0 | 2 | 5
Not Completed | 1 | 7 | 7
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Study Terminated by Sponsor | 1 | 6 | 6

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose, even if incomplete, of study treatment (TAK-580, TAK-202, or vedolizumab).
Groups:
- Arm 1: TAK-580 + Nivolumab: Participants in this group received TAK-580 400 mg, tablets, orally, once weekly along with nivolumab 3 mg/kg, infusion, intravenous, once every 2 weeks (up to Week 48).
- Total: Total of all reporting groups
Arm/Group | Arm 1: TAK-580 + Nivolumab | Arm 2: TAK-202 + Nivolumab | Arm 3: Vedolizumab + Ipilimumab + Nivolumab | Total
Number analyzed (Participants) | 1 | 9 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 | 63.9 (11.54) | 55.8 (16.36) | 58.5 (14.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 7 | 11
  Male | 0 | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 9 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 1 | 8 | 11 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 9 | 12 | 22
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 171.00 | 168.49 (10.479) | 170.00 (10.846) | 169.40 (10.170)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 77.80 | 77.42 (9.248) | 88.20 (26.786) | 83.32 (20.937)

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities (DLTs) During the Dose-escalation Safety Lead-in Phase
Description: DLTs was evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.
Time Frame: TAK-580 + Nivolumab and TAK-202 + Nivolumab: Baseline up to Week 9; Vedolizumab + Nivolumab + Ipilimumab: Baseline up to Week 7
Population: as for baseline characteristics
Measure: Number; unit: DLTs
Arm/Group | Arm 1: TAK-580 + Nivolumab | Arm 2: TAK-202 + Nivolumab | Arm 3: Vedolizumab + Ipilimumab + Nivolumab
Number analyzed (Participants) | 1 | 9 | 12
DLTs | 0 | 3 | 0

2. Secondary Outcome: Overall Response Rate (ORR) During the Dose-escalation Safety Lead-in Phase
Description: ORR based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. was the percentage of participants with complete response (CR) or partial response (PR). CR: was disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to less than (<) 10 millimeter (mm). PR: was at least a 30 percent (%) decrease in sum of diameter (SOD) of target lesions, taking as reference the baseline SOD.
Time Frame: Baseline up to Week 50
Population: Planned efficacy analyses was not performed as the study was terminated due to lack of enrollment, lack of clinical benefit and after the pre-specified stopping rule was met for diarrhea.
Arm/Group | Arm 1: TAK-580 + Nivolumab | Arm 2: TAK-202 + Nivolumab | Arm 3: Vedolizumab + Ipilimumab + Nivolumab
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Duration of Response (DOR) During the Dose-escalation Safety Lead-in Phase
Description: DOR based on RECIST version 1.1 was the time from the date of first documented confirmed CR/PR until the first documentation of confirmed progressive disease (PD) or death, whichever occurred first. CR: was disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to <10 mm. PR: at least 30% decrease in SOD of target lesions, taking as reference the baseline SOD persistence of one or more non- target lesions and/or maintenance of tumor marker level above the normal limits. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From date of first documented confirmed CR/PR until date of first documentation of PD or death (up to Week 50)
Population: as for outcome 2
Arm/Group | Arm 1: TAK-580 + Nivolumab | Arm 2: TAK-202 + Nivolumab | Arm 3: Vedolizumab + Ipilimumab + Nivolumab
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Progression-free Survival (PFS) During the Dose-escalation Safety Lead-in Phase
Description: PFS was the time from first dose date to date of the first documentation of confirmed PD or death, whichever occurred first. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions.
Time Frame: From first dose date to the date of the first documentation of confirmed PD or death (up to Week 50)
Population: as for outcome 2
Arm/Group | Arm 1: TAK-580 + Nivolumab | Arm 2: TAK-202 + Nivolumab | Arm 3: Vedolizumab + Ipilimumab + Nivolumab
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Overall Survival (OS) During the Dose-escalation Safety Lead-in Phase
Description: OS was the time from date of first dose of study drug until date of death from any cause.
Time Frame: From first dose of study drug until date of death from any cause (up to Week 50)
Population: as for outcome 2
Arm/Group | Arm 1: TAK-580 + Nivolumab | Arm 2: TAK-202 + Nivolumab | Arm 3: Vedolizumab + Ipilimumab + Nivolumab
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Reporting Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From the first dose of study drug up to 30 days after the last dose of study drug (up to Week 50)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Arm 1: TAK-580 + Nivolumab | Arm 2: TAK-202 + Nivolumab | Arm 3: Vedolizumab + Ipilimumab + Nivolumab
Number analyzed (Participants) | 1 | 9 | 12
participants
  TEAEs | 1 | 9 | 12
  SAEs | 1 | 2 | 7

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days (up to Week 50) after the last dose of study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Arm 1: TAK-580 + Nivolumab | Arm 2: TAK-202 + Nivolumab | Arm 3: Vedolizumab + Ipilimumab + Nivolumab
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/9 | 2/12
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/9 | 7/12
Other Adverse Events (participants affected / at risk) | 1/1 | 9/9 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: TAK-580 + Nivolumab (N=1) | Arm 2: TAK-202 + Nivolumab (N=9) | Arm 3: Vedolizumab + Ipilimumab + Nivolumab (N=12)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: TAK-580 + Nivolumab (N=1) | Arm 2: TAK-202 + Nivolumab (N=9) | Arm 3: Vedolizumab + Ipilimumab + Nivolumab (N=12)
Nausea (Gastrointestinal disorders) | 1 (3) | 6 (7) | 8 (10)
Fatigue (General disorders) | 1 (2) | 4 (8) | 9 (12)
Headache (Nervous system disorders) | 1 (1) | 3 (4) | 5 (10)
Pyrexia (General disorders) | 1 (1) | 3 (5) | 5 (9)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (5) | 5 (12)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (4) | 4 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 4 (4)
Hypothyroidism (Endocrine disorders) | 0 (0) | 4 (5) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 6 (10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 4 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (4) | 2 (4)
Chills (General disorders) | 0 (0) | 4 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (6) | 2 (3) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 3 (3)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Oropharyngeal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anorectal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bacterascites (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eosinophil percentage increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypohidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Micturition frequency decreased (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thyroid function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT02723006/Prot_SAP_000.pdf